CLINICAL TRIAL: NCT02430155
Title: Comparison of Condom-Loaded Foley's Catheter Versus Bakri Balloon for Treatment of Primary Postpartum Hemorrhage: A Randomized Controlled Trial
Brief Title: Balloon Tamponade for Atonic Primary Postpartum Hemorrhage
Acronym: UBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mamdouh Shaaban, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uterine balloon tamponade
Record Dates: First submitted 2015-03-24; First posted 2015-04-30 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Postpartum Hemorrhage
Keywords: condom-loaded Foley's catheter; Bakri balloon; primary atonic postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

ARMS (2):
- Bakri balloon group (Active Comparator): The women in this group will be managed by Bakri balloon
  Interventions: Device: Bakri balloon
- Condom loaded Foley's catheter group (Active Comparator): The women in this group will be managed by condom loaded Foley's catheter
  Interventions: Device: Condom loaded foley's catheter

INTERVENTIONS:
Device: Bakri balloon — is a 100% silicone construction, dual channel balloon catheter specifically designed and approved by FDA for intrauterine placement in cases of PPH. The Bakri balloon contains no latex, and therefore can be safely used in patients with latex allergies
  Arms: Bakri balloon group
Device: Condom loaded foley's catheter — Under aseptic precautions a sterile rubber catheter was inserted within the condom and tied near the mouth of the condom by a silk thread.
  Arms: Condom loaded Foley's catheter group

SUMMARY:
Postpartum hemorrhage (PPH) is responsible for around 25% of maternal mortality worldwide reaching as high as 60% in some countries.PPH can also be a cause of long-term severe morbidity, and approximately 12% of women who survive PPH will have severe anemia.

Postpartum hemorrhage has been defined as blood loss in excess of 500 ml in a vaginal birth and in excess of 1 L in a cesarean delivery.For clinical purposes, any blood loss that has the potential to produce hemodynamic instability should be considered a PPH. However, clinical estimates of blood loss are often inaccurate. Primary (immediate) PPH occurs within the first 24 hours after delivery and approximately 70% of these cases are due to uterine atony. Furthermore, uterine tony is defined as the failure of the uterus to contract adequately after the child is born.

Guidelines for the management of postpartum hemorrhage (PPH) involve a stepwise approach including the exclusion of retained products of conception and genital tract trauma. Uterine atony, which is the most common cause, the management of uterine atony is an established stepwise protocol that in many international guidelines.

Uterine massage is recommended for the treatment of PPH. Initiate uterine massages soon as excessive bleeding/uterine atony is identified. Intravenous oxytocin alone still is the recommended uterotonic drug for the treatment of PPH.

If intravenous oxytocin is unavailable or if the bleeding does not respond to oxytocin, intravenous ergometrine, oxytocin-ergometrine fixed dose or a prostaglandin drug (including sublingual misoprostol, 600 mcg) should be given. The use of intrauterine balloon tamponade is recommended for the treatment of primary PPH due to uterine atony in women who do not respond to uterotonics or if uterotonics are not available.

Since 1983, when Goldrath published evidence that inserting a Foley catheter in the uterus and inflating it with water could achieve tamponade, case series and other studies have suggested that various uterine balloon tamponade(UBT) devices may be effective in treating PPH. The studies used various types of UBT devices, including a condom catheter, a Foley catheter, the Sengstaken-Blakemore Esophageal Tube, the Rusch Balloon, and the Bakri Uterine Balloon. In 2007, a systematic review of treatment options for PPH found that 84% success rate of UBT does not significantly vary from surgical treatment outcomes.The World Health Organization (WHO), the International Federation of Gynecology and Obstetrics (FIGO), the American College of Obstetricians and Gynecologists(ACOG), the Royal College of Obstetricians and Gynecologists(RCOG), and the International Confederation of Midwives (ICM) recognize balloon tamponade as a method that could significantly improve the management intractable PPH, especially in low-resource areas.

In 2012, WHO updated the guidelines for the management of PPH and retained placenta to include: "The use of intrauterine balloon tamponade is recommended for the treatment of PPH due to uterine atony. This recommendation is now stronger than the previous guidelines. It can be used for women who do not respond to uterotonics or if uterotonics are not available. This procedure potentially can avoid surgery and is appropriate while awaiting transfer to a higher-level facility".Furthermore, FIGO included UBT as a recommended second-line intervention for the treatment of PPH in their updated guidelines issued in 2012.

Bakri first published the concept of intrauterine balloon technology in the management of hemorrhage secondary to placenta praevia-accreta during caesarean section with or without bilateral hypo gastric arterial ligation.In 2006, the ACOG Practice Bulletin, published by the American College of Obstetricians and Gynecologists, made mention of the Bakri postpartum balloon for its specifically tailored design that enables conservative management of uterine bleeding in cases of uterine atony and other causes of PPH.

The idea of using a condom as a balloon tamponade was first generated and evaluated in Bangladesh by Sayeba Akhter to fill a need and in response to the high cost of commercially available UBT devices.

ELIGIBILITY:
Inclusion Criteria:

* Women who accept to participate (either the patient or her first-kin if she is unconscious)
* Primary atonic postpartum hemorrhage

Exclusion Criteria:

* Traumatic postpartum hemorrhage
* With any suspected (e.g. prolonged rupture of membranes) or clinical evidence of infection
* Pre eclampsia.
* Diabetes mellietus(DM) with pregnancy
* History of Deep venous thrombosis (DVT) or other thromboembolic complication
* Rheumatic heart patients

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2016-03-04 (Actual)

PRIMARY OUTCOMES:
Number of patients who need surgical intervention to stop the bleeding | 1 year

SECONDARY OUTCOMES:
Time between insertion and stoppage of bleeding (minutes) | 1 year
Number of patients who need a blood transfusion | 1 year
Number of patients who developed fever | 1 year
The amount of blood loss (ml) after application of the balloon | 1 year
Number of patients who referred to Intensive care unit | 1 year
Number of patients who developed disseminated intravascular coagulopathy | 1 year
Duration (minutes) of bleeding after deflation of the balloon | 1 year
amount of bleeding (ml) after deflation of the balloon | 1 year

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374